CLINICAL TRIAL: NCT07006285
Title: T2 Biomarkers Predictive Value in Occupational Asthma After Cessation of Exposure.
Acronym: EAPT2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9224
Record Dates: First submitted 2024-11-08; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Asthma; Occupational Asthma; Occupational Diseases
MeSH Terms: conditions — Asthma; Asthma, Occupational; Occupational Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with occupational asthma (Other)
  Interventions: Other: Measure of T2 biomarkers

INTERVENTIONS:
Other: Measure of T2 biomarkers — T2 Biomarkers are estimated via induced sputum:
  Sputum is induced through increasing concentrations from 0.9 or 3% to 4% and 5% of hypertonic solution.
  Assessment of nonspecific bronchial hyperresponsiveness is realized by metacholine challenge

SUMMARY:
Occupational exposure is known to cause 15% of asthma cases. The main treatment for occupational asthma is to stop exposure if possible. Although, remission of occupational asthma only occurs in only 30 % of patients after cessation of exposure. There is currently no way of predicting which patients will go into remission after cessation of exposure.

In non-occupational asthma, the inflammatory biomarker T2 has allowed the entry into personalized medicine and can predict future exacerbations.

The investigators hypothesize that T2 biomarkers could be predictive markers for remission in occupational asthma after exposure cessation.

The investigators intend to carry out a follow-up study at the University Hospital of Strasbourg to perform the non-specific bronchial hyperresponsiveness test to assess remission in patients diagnosed with occupational asthma and to compare baseline T2 biomarkers in remission and non remission patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Diagnosis of occupational asthma by specific inhalation challenge
* Exposure to sensitizing agent avoided or reduced
* Able to understand the aims and risks of the research and to give free and informed consent
* For women of childbearing age: effective contraception in progress.
* Benefiting from social security coverage

Exclusion Criteria:

* Impossibility of giving the subject informed information (subject in emergency situation, difficulties in understanding the subject)
* Subject under court protection
* Subject under guardianship or curatorship
* Pregnant or breast-feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Remission of occupational asthma | Day 1
  Remission of occupational asthma is defined by absence of nonspecific bronchial hyperresponsiveness.
  Assessment of nonspecific bronchial hyperresponsiveness is realized by metacholine challenge
Comparison of TH2-type inflammation levels | Day 1
  To compare the level of Th2-type inflammation in sputum from patients in remission versus patients with persistent asthma.

SECONDARY OUTCOMES:
Remission of occupational rhinitis | Day 1
  Remission of occupational rhinitis is assessed by symptom score

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No